CLINICAL TRIAL: NCT02340624
Title: Optimizing Technology-Delivered Interventions for Smoking in Pregnancy: The Mommy Check-Up Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Elena Bronshtein, MFM Fellow, Wayne State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: WayneSU
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (8):
- Control group (No Intervention): No intervention(control group)
- condition 2 (Experimental): Intervention:Smokefreemoms texting
  Interventions: Behavioral: Referral to SmokeFreeMoms, Quitline or Brief intervention
- condition 3 (Experimental): Intervention: Quitline referral
  Interventions: Behavioral: Referral to SmokeFreeMoms, Quitline or Brief intervention
- condition 4 (Experimental): Intervention:Smokefreemoms texting and quitline referral
  Interventions: Behavioral: Referral to SmokeFreeMoms, Quitline or Brief intervention
- condition 5 (Experimental): Intervention: Brief intervention
  Interventions: Behavioral: Referral to SmokeFreeMoms, Quitline or Brief intervention
- condition 6 (Experimental): Intervention:Smokefreemoms texting and Brief intervention
  Interventions: Behavioral: Referral to SmokeFreeMoms, Quitline or Brief intervention
- condition 7 (Experimental): Intervention: Quitline referral and Brief intervention
  Interventions: Behavioral: Referral to SmokeFreeMoms, Quitline or Brief intervention
- condition 8 (Experimental): Intervention:Smokefreemoms texting, Quitline referral and Brief intervention
  Interventions: Behavioral: Referral to SmokeFreeMoms, Quitline or Brief intervention

INTERVENTIONS:
Behavioral: Referral to SmokeFreeMoms, Quitline or Brief intervention — 1. SmokeFreeMom is a mobile text messaging service designed for pregnant women across the United States to help them quit smoking. The program provides 24/7 encouragement, advice, and tips to help pregnant women and mothers quit smoking and stay quit.
  2. The 1-800 QuitLine provides smoking cessation services to Michigan residents who want to quit using tobacco. The Quit Line offers a personal health coach and participant toolkits to help tobacco users gain confidence and motivation they need to quit for good.
  3. Computer-delivered 5As (CD-5As) brief intervention The software platform to be used for this study features an interactive three-dimensional narrator, clear and relevant graphics, and aura;Participants use headphones for privacy while working with the computer.
  Arms: condition 2; condition 3; condition 4; condition 5; condition 6; condition 7; condition 8

SUMMARY:
Tobacco smoking in pregnancy remains one of the most important and preventable cause of adverse pregnancy outcomes. Data from National Survey of Drug Use and Health (NSDUH) suggests, that the annual average rates of current cigarette use among women aged 15 to 44 who were not pregnant decreased from 30.7 percent in 2002-2003 to 24.0 percent in 2012-2013. However, the prevalence of cigarette use among pregnant women in this age range did not change significantly during the same time period (18.0 percent in 2002-2003 and 15.4 percent in 2012-2013)Smoking cigarettes during pregnancy and nursing causes considerable health damage to the fetus and to the infant during the initial growth phase. An estimated 19.8 million women in the United States smoke. Nationally, 23 percent of women report smoking in the 3 months before pregnancy, while 13 percent report smoking in the last 3 months of pregnancy. Overwhelming evidence suggests that maternal smoking during pregnancy is associated with an adverse pregnancy outcomes including IUGR, placenta previa, abruption placentae, preterm premature rupture of membranes, low birth weight, perinatal mortality, intrapartum stillbirth and ectopic pregnancy. Moreover, prenatal exposure to tobacco smoke also increases risk of attention deficit and hyperactivity disorder (ADHD) and sudden infant death syndrome (SIDS) in the offspring.Children born to mothers who smoke during pregnancy are at increased risk of asthma, infantile colic, and childhood obesity.

Brief interventions are shown to be associated with small but clear increases in smoking cessation in pregnancy, but are rarely used. Technology may fill this void. For the present study, pregnant women reporting smoking during pregnancy will be recruited and randomly assigned to one of eight combinations of three technology-delivered intervention approaches: Brief intervention, Quitline referral, and "SmokeFreeMoms" text messages (http://women.smokefree.gov/smokefreemom.aspx).

DETAILED DESCRIPTION:
The study will be introduced to pregnant smokers age 18-45 by clinic staff at the DMC prenatal care clinic located at the University Health Center, or at a UPG prenatal care clinic. Medical staff will give potential participants a flyer briefly describing the study and providing a link to a website (www.mommycheckup.net). Participants who meet all inclusions and exclusion criteria and pass the quiz will be randomized to one of the eight possible combinations of the three different interventions: Brief intervention, SmokeFreeMoms texting, or Quitline referral. This use of a factorial design to examine the relative efficacy of various intervention components is consistent with the Multiphase Optimization Strategy (the MOST) approach. Follow-up evaluation will take place at 4 weeks, and will have two elements, one computer- or mobile device-based and the other involving provision of a saliva/urine and breath sample. These will be done separately (if the participant does the online version remotely) or together (if the participant does the online component while providing the samples). Online follow-up: Participants will be sent a link to the online system, through which they will be asked about smoking. The clinic follow-up assessment will be performed at the next clinic visit. All participants will be asked to provide a urine sample (to be tested for cotinine, a biomarker of cigarette smoking) and a breath sample (to be tested for carbon monoxide level).

Data will be analyzed using a 2 (brief intervention yes vs. no)) X 2 (texting referral yes-no) X 2 (quitline referral yes-no) ANCOVA (controlling for baseline smoking) test with a power of 75%, α=0.05, and 200 patients will be required for this study. The information will be analyzed using SPSS. We will examine main effects for each of the three factors. Based on an incidence of tobacco smoke in pregnancy, the total recruitment will take 3-4 months.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18-45, at less than 30 weeks gestation, who smoke daily, have access to a mobile device and are willing to accept text messages.

Exclusion Criteria:

* not having access to a mobile device with a texting plan.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-04 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Abstinence from smoking | Seven-day point-prevalence
  To compare the effects on smoking of an online brief intervention to those of referral to a free online text messaging intervention, and to those of free phone counseling through the Michigan Quitline.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sokol, MD, Study Director — WSU
Locations (1):
- DMC, Detroit, Michigan, United States

REFERENCES:
- [Background] Kleijer ME, Dekker GA, Heard AR. Risk factors for intrauterine growth restriction in a socio-economically disadvantaged region. J Matern Fetal Neonatal Med. 2005 Jul;18(1):23-30. doi: 10.1080/14767050500127674. PMID 16105788